CLINICAL TRIAL: NCT02018237
Title: The Effect of High Fructose Corn Syrup Feeding in Nonalcoholic Fatty Liver Disease
Brief Title: High Fructose Corn Syrup
Acronym: Fructose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-12111
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Nonalcoholic Fatty Liver Disease; Obesity
Keywords: Obesity; Nonalcoholic fatty liver disease; High fructose corn syrup
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity | interventions — High Fructose Corn Syrup

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAFLD (Active Comparator): Subjects with nonalcoholic fatty liver disease (NAFLD) will complete baseline testing and then be assigned to either the high fructose corn syrup diet or the standard diet (low in high fructose corn syrup) for 4 weeks. Post intervention testing will be completed after the subjects have completed the 4 week diet intervention.
  Interventions: Behavioral: High fructose corn syrup diet; Behavioral: Standard diet (low in high fructose corn syrup)
- Non-NAFLD (Active Comparator): Subjects without nonalcoholic fatty liver disease (Non-NAFLD) will complete baseline testing and then be fed a high fructose corn syrup diet for 4 weeks. Post intervention testing will be completed after the subjects have completed the 4 week diet intervention.
  Interventions: Behavioral: High fructose corn syrup diet

INTERVENTIONS:
Behavioral: High fructose corn syrup diet — Subjects will consume a high fructose corn syrup diet for 4 weeks. The food will be prepared by the bio-nutrition kitchen, and meals will be picked up every 3-4 days.
Behavioral: Standard diet (low in high fructose corn syrup) — Subjects will consume a standard diet (low in high fructose corn syrup) for 4 weeks. The food will be prepared by the bio-nutrition kitchen, and meals will be picked up every 3-4 days.
  Arms: NAFLD

SUMMARY:
The purpose of this research study is to learn more about how high fructose corn syrup, a sugar used to sweeten drinks and foods, affects metabolism in obese persons with and without nonalcoholic fatty liver disease. Eligible participants will be studied before and after eating a diet high in high fructose corn syrup or a standard diet (low in high fructose corn syrup) for four weeks.

ELIGIBILITY:
Inclusion Criteria:

* IHTG >6.5% or <5%
* BMI 30.0-45.0 kg/m²
* Sedentary
* Consume <10% calories from high fructose corn syrup
* Weight stable for previous 3 months

Exclusion Criteria:

* IHTG 5.1-7.9%
* Children
* Adults over 65 years
* Pregnant
* Lactating
* Exercise >1.5 hours/week
* Hepatitis B or C
* Diabetes
* History of liver disease
* History of alcohol abuse
* Severe hypertriglyceridemia (>300 mg/dl)
* Smokers
* Anemia (Hemoglobin <10mg/dl)
* Not weight stable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in intrahepatic triglyceride (IHTG) content | 4 weeks
  Determine the effect of 4-week isocaloric diet high in high fructose corn syrup (HFCS) on IHTG content measured by magnetic resonance spectroscopy (MRS).
Hepatic lipid metabolism | 4 weeks
  Determine the effect of 4-week isocaloric diet high in HFCS on hepatic lipid metabolism [de novo lipogenesis, very low density lipoprotein-triglyceride (VLDL-TG) and very low density lipoprotein-Apolipoprotein B100 (VLDL-ApoB) secretion rates] by using stable isotope tracer methods.
Multi-organ insulin sensitivity | 4 weeks
  Determine the effect of 4-week isocaloric diet high in HFCS on multi-organ insulin sensitivity by using a one stage hyperinsulinemic euglycemic clamp procedure in conjunction with muscle and adipose tissue biopsies.
Uric acid metabolism | 4 weeks
  Determine the effect of 4-week isocaloric diet high in HFCS on uric acid metabolism by measuring post-prandial serum uric acid concentrations and using stable isotope tracer method.

CONTACTS AND LOCATIONS:
Overall Officials: Shelby A Sullivan, MD, Principal Investigator — Associate Professor of Medicine; Samuel Klein, MD, Principal Investigator — Professor of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States